CLINICAL TRIAL: NCT06081777
Title: A Study Evaluating MRD Biomarker in Patients With Potentially Resectable Stage III Non-small Cell Lung Cancer
Brief Title: Significance of MRD Monitoring in Patients With Potentially Resectable Stage III Non-small Cell Lung Cancer
Acronym: MRDinS3LC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: LGH2022144
Record Dates: First submitted 2023-06-24; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: NSCLC
Keywords: MRD, potentially resectable NSCLC, stage III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — 1. To evaluate the consistency of node MRD results with cCR(clinical imaging) and its relationship with pCR/non-pCR after neoadjuvant therapy;
  2. To evaluate the relationship between baseline MRD results and prognosis, and to evaluate the relationship between multi-node MRD results and prognosis during follow-up;
  3. Good/bad prognosis of adjuvant therapy and baseline mutant spectrum analysis, baseline ctDNA frequency analysis, pCR results analysis;
  4. An exploratory analysis was conducted on the relationship between negative MRD and survival between patients who received surgery and those who did not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arms1：For stage III NSCLC patients who underwent complete resection.: Immunotherapy alone or chemotherapy combined with immunotherapy. Collect patients' baseline puncture tissues, peripheral blood samples from multiple nodes after new adjuvant treatment, surgery (if any), adjuvant treatment, and follow-up, and carry out for 1021-MRD analysis through tumor-informed personalized monitoring MRD test kit.
  Assigned Interventions：1021-MRD analysis
- Arms 2：For stage III NSCLC patients who underwent concurrent radio-chemotherapy.: Immunotherapy alone or chemotherapy combined with immunotherapy. Collect patients' baseline puncture tissues, peripheral blood samples from multiple nodes after new adjuvant treatment, surgery, adjuvant treatment, and follow-up, and carry out for 1021-MRD analysis through tumor-informed personalized monitoring MRD test kit.
  Assigned Interventions：1021-MRD analysis

SUMMARY:
Stratification of postoperative ctDNA status can effectively assess the risk of recurrence in patients. In addition, the multi-node dynamic monitoring of ctDNA is more effective in predicting the recurrence risk of patients. In this study, EGFR/ALK negative potentially resectable Stage III non-small cell lung cancer were enrolled. Baseline tissues, Peripheral blood samples of patients at baseline puncture tissue, after neoadjuvant therapy, after surgery (if any), after adjuvant therapy, and at multiple nodes during follow-up were collected for 1021-MRD analysis through tumor-informed personalized monitoring MRD test kit. This study aim to explore MRD biomarker in patients with potentially resectable stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
In this prospective study, 65 patients with potentially operable non-small cell lung cancer without driving gene EGFR/ALK mutation in stage III were enrolled in this prospective study. peripheral blood samples from multiple nodes after neoadjuvant therapy, postoperative (if any), adjuvant therapy and follow-up were collected and analyzed by high-throughput sequencing in the target region. Patients were enrolled in the study for 1 year, followed up for 2 years, and the study lasted for 3 years. The patients were followed up for 2 years according to the standard diagnosis and treatment path, with a total of 9 times of follow-up, all of which were 3-month follow-up plan of the standard diagnosis and treatment path, and the follow-up examination was conducted in accordance with clinical standards.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, age ≥ 18 and ≤ 80.
2. patients with stage Ⅲ non-small cell lung cancer confirmed by histology or cytology have potential surgical opportunities.
3. No driving gene EGFR/ALK mutation.
4. PS = 0-1.
5. the treatment process cooperated with the provision of clinicopathological and imaging data needed in the research process, followed up and collected the blood of the clinical efficacy evaluation nodes, and agreed to use the test data for follow-up research and product development.

Exclusion Criteria:

1. patients suffering from other malignant tumors.
2. patients change the treatment regimen before receiving the specified treatment or before the disease progresses.
3. Patients could not cooperate with the study for follow-up according to the defined clinical follow-up period;
4. Patients were unable to accept or provide imaging and other designated therapeutic evaluation means.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Capable of giving signed informed consent, age ≥ 18 and ≤ 80.
  2. patients with stage Ⅲ non-small cell lung cancer confirmed by histology or cytology have potential surgical opportunities.
  3. No driving gene EGFR/ALK mutation.
  4. PS = 0-1.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (RECIST) | follow-up time: 2 years
  Disease-free survival (RECIST)： the survival time from operation or radiation to recurrence

SECONDARY OUTCOMES:
OS | follow-up for 2 years
  overall survival from the enrollment to death
The prediction of recurrence by positive MRD | follow-up for 2 years
  Whether the prediction of recurrence by positive MRD is earlier than that confirmed by clinical diagnosis.
pCR rate of MRD-negative patient | 2 years
  pCR rate of MRD-negative patient
Negative MRD rate in pCR patients | follow-up time: 2 years
  Negative MRD rate in pCR patients
2-year DFS of ctDNA-negative patients in operation group / inoperable group | follow-up time: 2 years
  2-year DFS of ctDNA-negative patients in operation group / inoperable group

CONTACTS AND LOCATIONS:
Overall Officials: Yuyan Wang, doctorate, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Yuyan Wang, Beijing, China

IPD SHARING:
Plan to Share IPD: No